CLINICAL TRIAL: NCT00655850
Title: Pilot Phase II Study of Metronomic Chemotherapy in Combination With Avastin in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Lower Dose Chemotherapy Given More Frequent With Avastin to Treat Advanced Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F070727010; UAB 0709
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; Metronomic Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Paclitaxel; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel and Gemcitabine + Avastin (Experimental): Patients will be treated with metronomic chemotherapy with paclitaxel and gemcitabine weekly for 3 out of 4 weeks which constitutes one cycle (4 weeks). Avastin will be administered every 2 weeks. Treatment with metronomic chemotherapy and Avastin will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity, or withdrawal of consent. Maintenance therapy with Avastin will continue until disease progression, intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine; Biological: Avastin

INTERVENTIONS:
Drug: Paclitaxel — * Prior to receiving paclitaxel, all patients will receive the following premedications one hour before the infusion:
  * Dexamethasone 20mg, intravenously (IV)
  * Diphenhydramine 50 mg IV
  * Ranitidine 50 mg IV
  * Paclitaxel will be administered after the gemcitabine infusion as a 1 hour (IV) infusion.
  * The initial dose of paclitaxel is 80 mg/m2/weekly for 3 out of 4 weeks (Day 1, 8, 15)
  Paclitaxel Dose Levels:
  * Dose Level 1 ________80 mg/m2/weekly
  * Dose Level -1 ________70 mg/m2/weekly
  Other Names: Taxol
Drug: Gemcitabine — Premedication
  * Prophylactic antiemetics: 5-HT3-receptor antagonist prior to infusion with gemcitabine.
  * Prior to receiving paclitaxel chemotherapy
  * Gemcitabine will be given at the initial dose of 200mg/m2/week (Dose Level 1) for 3 out of 4 weeks (Day 1, 8, 15), as a 30 minute (IV) infusion.
  * The dose of gemcitabine can be escalated to 300mg/m2/weekly (Dose Level 2) after the first cycle of treatment if no significant toxicity is experienced.
  Gemcitabine Dose Levels:
  * Dose Level 2 ________300 mg/m2/weekly
  * Dose Level 1 ________200 mg/m2/weekly
  * Dose Level -1 ________150 mg/m2/weekly
  Other Names: Gemzar
Biological: Avastin — * The dose of Avastin is 10 mg/kg IV every 2 weeks
  * It will be administered following the administration of chemotherapy
  * The first infusion will be administered over 90 minutes; if well tolerated, the second and subsequent doses will be administered as a 60-minute and 30-minute infusion, respectively.
  * It should not be administered or mixed with dextrose solutions.
  Other Names: Anti-VEGF

SUMMARY:
This study is being done to determine the overall progression-free survival (PFS) in patients with advanced or metastatic (Stage IIIB - pleural effusion/IV), non-squamous histology NSCLC treated with metronomic chemotherapy plus Avastin. Also, currently there are no defined markers that predict for clinical benefit to Avastin. Preliminary studies show that there are several observations that support the concept of metronomic chemotherapy with or without the combination of an anti-angiogenic agent. The metronomic chemotherapy with Avastin was shown to enhance the clinical endpoints of the study (response rate and progressive-free survival). Proof of metronomic scheduling requires the development of appropriate intermediate surrogate markers. Several markers will be assessed.

DETAILED DESCRIPTION:
This is a non-randomized, open-label, pilot Phase II study of metronomic chemotherapy plus Avastin in chemo naïve subjects with advanced non-squamous, non-small cell carcinoma of the lung. The primary endpoint of this study is to assess the overall progression-free survival.

Subjects will be treated with metronomic chemotherapy with paclitaxel and gemcitabine weekly for 3 out of 4 weeks, and Avastin will be administered every 2 weeks. Treatment with metronomic chemotherapy will be expressed as a 4-week cycle. Tumor response to treatment will be evaluated every 8 weeks.

Treatment with metronomic chemotherapy and Avastin will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity, or withdrawal of consent. Maintenance therapy with Avastin will then continue until disease progression, intolerable toxicity or withdrawal of consent.

Potential biologic parameters to monitor anti-tumor activity of metronomic chemotherapy will be evaluated in 10 subjects. These biomarkers include: sequential determination of blood levels of VEGF, VEGFR2, thrombospondin-1, E-selectin, ICAM-1, and circulating endothelial cells and endothelial precursor cells.

ELIGIBILITY:
Inclusion Neutrophil Count greater than or equal to 1500/μL

* Platelet Count greater than or equal to 100,000/μL
* Hemoglobin greater than or equal to 9.0g/dL
* Total Bilirubin ≤ 1.5mg/dL
* Transaminases ≤ 2.5 x ULN
* Serum Creatinine ≤ 1.5 x ULN
* Proteinuria: Urine protein: creatinine (UPC) ratio < 1.0 at screening OR Urine dipstick for proteinuria < 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).

INR ≤ 1.5 and a PTT no greater than the ULN

* Subjects must be 19 years or older.
* Subjects with a history of hypertension must be well-controlled (< 150/100) on a stable regimen of anti-hypertensive therapy.
* Subjects must not have serious non-healing wound ulcer, or bone fracture, or major surgical procedure within 28 days prior to starting treatment.
* Subjects must not have radiation therapy within 3 weeks prior to initiation of treatment.
* Female subjects must be postmenopausal, surgically sterile, or using effective contraception. All females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the initiation of treatment.
* Informed consent must be obtained in writing prior to the initiation of treatment.

Exclusion Criteria

* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last five years

Avastin-Specific Exclusions

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known CNS disease, except for treated brain metastasis Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (greater than or equal to 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio greater than or equal to 1.0 at screening
* Known hypersensitivity Criteria:
* Pathological-proven NSCLC except squamous cell carcinoma as the predominant histology.
* Advanced NSCLC: Stage IIIB with pleural effusion or Stage IV or recurrent disease.
* Measurable or non-measurable disease as defined by solid tumor response criteria (RECIST)
* ECOG Performance Status 0 to 1.
* No prior systemic chemotherapy or biologic therapy.
* Required laboratories (obtained ≤ 1 week prior to the initiation of treatment)
* Absolutely any component of Avastin
* Pregnancy (positive pregnancy test) or lactation. Use of effective means of contraception (men and women) in patients of child-bearing potential
* Intrathoracic lung carcinoma of squamous cell histology Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is acceptable. Patients with extrathoracic-only squamous cell NSCLC are eligible. Patients with only peripheral lung lesions (of any NSCLC histology) will also be eligible (a peripheral lesion is defined as a lesion in which the epicenter of the tumor is less than or equal to 2 cm from the costal or diaphragmatic pleura in a three-dimensional orientation based on each lobe of the lung and is greater than 2 cm from the trachea, main, and lobar bronchi).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-03; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: March 2008, Primary Completion Date: September 2015 and Study Completion Date: September 2016. Recruitment location: University of Alabama at Birmingham.
Pre-assignment Details: This study is being done to determine the overall progression-free survival (PFS) in patients with advanced or metastatic (Stage IIIB - pleural effusion/IV), non-squamous histology Non-Small Cell Lung Cancer (NSCLC) treated with metronomic chemotherapy plus Avastin.
Groups:
- Paclitaxel and Gemcitabine + Avastin: Patients will be treated with metronomic chemotherapy with paclitaxel and gemcitabine weekly for 3 out of 4 weeks which constitutes one cycle (4 weeks). Avastin will be administered every 2 weeks. Treatment with metronomic chemotherapy and Avastin will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity, or withdrawal of consent. Maintenance therapy with Avastin will continue until disease progression, intolerable toxicity, or withdrawal of consent.
  Paclitaxel: -Prior to receiving paclitaxel, all patients will receive the following premedications one hour before the infusion:
  * Dexamethasone 20mg, intravenously (IV)
  * Diphenhydramine 50 mg IV
  * Ranitidine 50 mg IV
  * Paclitaxel will be administered after the gemcitabine infusion as a 1 hour (IV) infusion
  * The initial dose of paclitaxel is 80 mg/m2/weekly for 3 out of 4 weeks (Day 1, 8, 15)
  Paclitaxel Dose Levels:
  * Dose Level 1 ________80 mg/m2/weekly
  * Dose Level -1 _____
Period: Overall Study
Arm/Group | Paclitaxel and Gemcitabine + Avastin
Started | 39
Completed | 36
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patients were required to be over 18 years of age, have stage IV, histologically proven non-squamous NSCLC, have Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1, have received no prior systemic therapy for cancer, and have adequate organ function.
Arm/Group | Paclitaxel and Gemcitabine + Avastin
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 59.5 [37 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression Free Survival is defined as the number of days from the day the subject started treatment to the day the subject experiences disease progression in accordance with the Response Evaluation Criteria Solid Tumors (RECIST v1.0). The RECIST criteria indicates progression as a 20% increase in the total tumor measurement over nadir value or the appearance of new lesions.
Time Frame: Baseline to 24 months
Population: Participants with advanced chemotherapy naïve with non-squamous non-small cell lung cancer.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel and Gemcitabine + Avastin
Number analyzed (Participants) | 36
months | 8.5 [5 to 10]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: All adverse events will be recorded as to the grade and relationship to the study drug in accordance with the Common Terminology Criteria for Adverse Events (CTCAE v 3.0)
Time Frame: Baseline through duration of treatment an average of 1 year
Population: Participants with advanced chemotherapy naïve with non-squamous non-small cell lung cancer.
Measure: Number; unit: participants
Arm/Group | Paclitaxel and Gemcitabine + Avastin
Number analyzed (Participants) | 36
participants | 36

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the number of days from the day the subject started treatment to the day the subject experiences death or lost to follow up.
Time Frame: Baseline up to 84 months
Population: Participants with advanced chemotherapy naïve with non-squamous non-small cell lung cancer.
Measure: Median (Full Range); unit: months
Groups:
- Paclitaxel and Gemcitabine + Avastin: Patients will be treated with metronomic chemotherapy with paclitaxel and gemcitabine weekly for 3 out of 4 weeks which constitutes one cycle (4 weeks). Avastin will be administered every 2 weeks. Treatment with metronomic chemotherapy and Avastin will continue for a total of 6 cycles unless there is evidence of disease progression, intolerable toxicity, or withdrawal of consent. Maintenance therapy with Avastin will continue until disease progression, intolerable toxicity, or withdrawal of consent
  Paclitaxel: -Prior to receiving paclitaxel, all patients will receive the following premedications one hour before the infusion:
  * Dexamethasone 20mg, intravenously (IV)
  * Diphenhydramine 50 mg IV
  * Ranitidine 50 mg IV
  * Paclitaxel will be administered after the gemcitabine infusion as a 1 hour (IV) infusion.
  * The initial dose of paclitaxel is 80 mg/m2/weekly for 3 out of 4 weeks (Day 1, 8, 15)
  Paclitaxel Dose Levels:
  * Dose Level 1 ________80 mg/m2/weekly
  * Dose Level -1 _____
Arm/Group | Paclitaxel and Gemcitabine + Avastin
Number analyzed (Participants) | 36
months | 25.5 [15 to 35]

4. Secondary Outcome: Objective Response Rate
Description: The percentage of patients who achieve a complete response and partial response according to RECIST criteria (v1.0).
Time Frame: Baseline up to 12 months
Population: Participants with advanced chemotherapy naïve with non-squamous non-small cell lung cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel and Gemcitabine + Avastin
Number analyzed (Participants) | 36
Participants | 22

ADVERSE EVENTS:
Time Frame: Baseline up to 24 months
Arm/Group | Paclitaxel and Gemcitabine + Avastin
All-Cause Mortality (participants affected / at risk) | 2/36
Serious Adverse Events (participants affected / at risk) | 25/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and Gemcitabine + Avastin (N=36)
Neutropenia: Induction (Blood and lymphatic system disorders) | 6 (6)
Fatigue: Induction (General disorders) | 1 (1)
Nausea Vomiting: Induction (Gastrointestinal disorders) | 1 (1)
Hypertension Grade: end of Cycle 1 (Cardiac disorders) | 1 (1)
Hypertension: end of induction (Cardiac disorders) | 5 (5)
Hypertension grade: maintenance (Cardiac disorders) | 4 (4)
Proteinuria: Induction (Renal and urinary disorders) | 4 (4)
Proteinuria: Maintenance (Renal and urinary disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and Gemcitabine + Avastin (N=36)
Neutropenia: Induction (Blood and lymphatic system disorders) | 14 (14)
Thrombocytopenia: Induction (Blood and lymphatic system disorders) | 17 (17)
Anemia: Induction (Blood and lymphatic system disorders) | 27 (27)
Nausea/Vomiting: Induction (Gastrointestinal disorders) | 17 (17)
Diarrhea: Induction (Gastrointestinal disorders) | 20 (20)
Fatigue: Induction (General disorders) | 32 (32)
Neuropathy: Induction (Nervous system disorders) | 19 (19)
Hypertension grade: end of Cycle 1 (Cardiac disorders) | 26 (26)
Hypertension grade: end of induction (Cardiac disorders) | 32 (32)
Hypertension grade: maintenance (Cardiac disorders) | 17 (17)
Proteinuria: Induction (Renal and urinary disorders) | 14 (14)
Proteinuria: Maintenance (Cardiac disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No